CLINICAL TRIAL: NCT07260058
Title: Clinical Study on the Safety and Efficacy of Autologous Immune Cell Therapy for Advanced Solid Tumors
Brief Title: Immune Cell Therapy for Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Liaoning Medical Diagnosis and Treatment Technology Research and Development Co., Ltd. (Industry)
Collaborators: Liaoning Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LNMDTC-Solid tumor
Record Dates: First submitted 2025-09-28; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer (Locally Advanced or Metastatic); Liver Cancer (Locally Advanced or Metastatic); Colorectal Cancer (Locally Advanced or Metastatic); Breast Cancer (Locally Advanced or Metastatic); Advanced Solid Tumors
Keywords: Advanced Solid Tumors; Metastatic Lung Cancer; Metastatic Liver Cancer; Metastatic Colorectal Cancer; Metastatic Breast Cancer; Autologous Immune Cell Therapy; Dendritic Cell Vaccine; CIK Cells; NK Cells
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Liver Neoplasms; Colorectal Neoplasms; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This study employs a sequential, two-phase design that incorporates both non-randomized and randomized components:
  Phase I (Safety Lead-in): This initial phase is a non-randomized, biomarker-directed study. Participants are assigned to one of two autologous immune cell therapy regimens based on their HLA-A phenotype:
  HLA-A positive participants receive DC-CIK therapy.
  HLA-A negative participants receive NK cell therapy. The primary objective of this phase is to evaluate the safety and feasibility of the cell products.
  Phase II (Expansion): This subsequent phase is a randomized, parallel-group, controlled study. Following the HLA-A stratification:
  HLA-A positive participants are randomized to either the DC-CIK + Chemotherapy group or the Chemotherapy alone group.
  HLA-A negative participants are randomized to either the NK + Chemotherapy group or the Chemotherapy alone group.
  The primary objective of this phase is to evaluate the efficacy (Objective Response Rate) of the combinatio
Masking Description: This is an open-label study where no masking (blinding) is used. The nature of the interventions makes masking infeasible. Participants, care providers, investigators, and outcomes assessors will all be aware of the treatment group assignments.
  The key reasons for the open-label design are:
  Distinct Procedures: The autologous immune cell therapy requires a specific process of leukapheresis (blood draw) for cell manufacturing, which is not required for participants in the chemotherapy-only control groups.
  Different Administration Routes: The dendritic cells (DC) are administered via subcutaneous injection, while the CIK and NK cells are administered via intravenous infusion. These routes and the appearance of the cell products differ visibly from standard intravenous chemotherapy.
  Lack of Placebo: The study protocol does not include the manufacture of a matched placebo for the cellular products to mimic the appearance and administration process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): This arm includes all participants who receive the investigational autologous immune cell therapy (either DC-CIK or NK cells), either alone or in combination with chemotherapy. It consolidates the following original arms:
  Phase I - DC-CIK Therapy Arm Intervention Name: Autologous DC-CIK Cells
  Phase I - NK Therapy Arm Intervention Name: Autologous NK Cells
  Phase II - DC-CIK + Chemotherapy Arm Intervention Name: Autologous DC-CIK Cells+Standard Chemotherapy
  Phase II - NK + Chemotherapy Arm Intervention Name:Autologous NK Cells+Standard Chemotherapy
  Interventions: Biological: Autologous immune Cells; Drug: Standard chemotherapy
- Control Group (Active Comparator): This arm includes all participants who receive standard chemotherapy alone, without any investigational cell therapy. It consolidates the following original arms:
  Phase II - Chemotherapy Control Arm (HLA-A Positive)
  Phase II - Chemotherapy Control Arm (HLA-A Negative)
  Interventions: Drug: Standard chemotherapy

INTERVENTIONS:
Biological: Autologous immune Cells — 1. Autologous DC-CIK Cells：Dendritic Cells (DC) and Cytokine-Induced Killer (CIK) cells are manufactured ex vivo from the participant's own peripheral blood mononuclear cells (PBMCs). DC cells (>5x10⁶ cells) are administered via subcutaneous injection. CIK cells (>5x10⁹ cells) are administered via intravenous infusion.
  2. Autologous NK Cells：Natural Killer (NK) cells are manufactured ex vivo from the participant's own peripheral blood mononuclear cells (PBMCs). NK cells (≥3x10⁹ cells) are administered via intravenous infusion.
  Arms: Experimental Group
Drug: Standard chemotherapy — Investigator's choice of standard chemotherapy regimen(s) appropriate for the participant's specific type of advanced solid tumor (lung, liver, colorectal, or breast cancer), administered according to local clinical practice.

SUMMARY:
The autologous immune cell induction technology used in this project involves transforming peripheral blood mononuclear cells (PBMC) into autologous DC cells, NK cells, CIK cells and other immune cells through cytokine induction, and then re-administering them to the patients. This therapy utilizes biotechnology to culture the immune cells of cancer patients in vitro and then re-infuse them back into the body, stimulating and enhancing the body's own immune function, killing and inhibiting cancer cells, eliminating small and residual lesions, or achieving the goal of treating cancer by significantly inhibiting the proliferation of residual cancer cells.

DETAILED DESCRIPTION:
This project focuses on the DC autologous immunocyte therapy based on the core technology of screening tumor antigen dominant CTL epitope peptides through independent patent technology. It is a cutting-edge research direction in the field of tumor immunotherapy in recent years. The non-engineered DC cells induced by special induction techniques can effectively overcome the shortcomings of the poor therapeutic effect of engineered gene editing technology on solid tumors, and effectively achieve targeted killing of tumors. The DC-CIK immunocyte therapy adopted in this project utilizes the original discovery of HLA-A molecule-restricted tumor-related antigen CTL epitope peptides to modify DC. On the one hand, through subcutaneous injection in vivo, it induces CD8+ T cells to produce CTL with memory function to play a role in eliminating and monitoring the protein with high expression of the tumor antigen source. On the other hand, it induces CD8+ T cells to produce CTL with memory function in vitro, and directly reinfuses CTL to exert the role of eliminating and monitoring the protein with high expression of the tumor antigen source. In the previous experimental studies, the CTL induced by G22 antigen-loaded DC has shown significant "identification" and targeted "killing" capabilities against various solid tumor cell lines and primary tumor cells isolated from tumor tissues. In animal experiments, it also shows the ability to induce the body to produce a strong immune response against various solid tumors such as breast cancer and non-small cell lung cancer, significantly inhibiting tumor growth, prolonging progression-free survival, and showing no obvious toxic side effects, having a promising application prospect. It has high individualization: customized based on the tumor mutation spectrum of patients, avoiding "off-target" damage to normal tissues. It has high safety: clinical studies have shown that the side effects are mild, mainly including injection site reactions or transient fever 37. Combined treatment potential: it can be used in combination with PD-1 inhibitors, chemotherapy or radiotherapy to enhance efficacy.

At present, self-active immune cell therapy based on tumor antigen-specific CTL epitope peptides has achieved significant progress in both research and clinical application in China. Personalized tumor vaccines, targeted immunoregulatory strategies for the tumor microenvironment, and combination treatment strategies are providing new concepts and methods for tumor therapy. In summary, the "Clinical Research on Safety and Effectiveness of Autologous Immune Cell Therapy for Advanced Solid Tumors" is expected to provide a clinical trial basis for the development of safe and effective clinical immunotherapies for patients with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, an individual must meet all of the following criteria:

1. The participant must voluntarily participate in the study and provide written informed consent。
2. Age ≥ 18 years, male or female.
3. Histologically and/or cytologically confirmed locally advanced or metastatic solid tumor: lung cancer, liver cancer, colorectal cancer, or breast cancer.
4. ECOG (Eastern Cooperative Oncology Group) performance status score ≤ 2.
5. Life expectancy ≥ 3 months.
6. Has not received any other cellular immunotherapy within 3 months prior to enrollment.
7. Has at least one measurable lesion according to RECIST (Response Evaluation Criteria in Solid Tumors) Version 1.1.
8. Adequate organ function, defined as follows:

Hematology:

White Blood Cell (WBC) count > 3.5 × 10⁹/L Lymphocyte count > 0.9 × 10⁹/L Monocyte count > 0.16 × 10⁹/L Absolute Neutrophil Count (ANC) > 1.5 × 10⁹/L Platelet (PLT) count > 75 × 10⁹/L Hemoglobin (HB) > 75 g/L Blood Biochemistry： Total bilirubin ≤ 1.5 × ULN (Upper Limit of Normal) Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 2.5 × ULN (≤ 5 × ULN if liver metastases are present)

Coagulation:

Prothrombin Time (PT) and International Normalized Ratio (INR) ≤ 1.5 × ULN

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Prior receipt of any salvage chemotherapy, implanted intraperitoneal chemotherapy, targeted therapy, or biological immunotherapy (except: patients whose disease progressed more than 6 months after completing adjuvant, neoadjuvant, or radiosensitizing chemotherapy, or more than 1 month after intraperitoneal chemoperfusion/wash, are eligible, provided chemotherapy-related toxicities have recovered to Grade 1 or below, excluding alopecia).
2. Major surgical procedure within 4 weeks prior to enrollment, with incomplete recovery from side effects.
3. History of any active malignancy within 5 years, except for the specific cancer under investigation in this trial and cured localized tumors such as carcinoma in situ of the cervix, basal cell carcinoma of the skin, and prostate carcinoma in situ.
4. Presence of more than a small amount of pericardial effusion, or uncontrolled pleural or peritoneal effusion, defined as: detectable by physical examination at screening, or requiring therapeutic paracentesis during the screening period.
5. Inability to tolerate peripheral blood collection due to various reasons (e.g., severe coronary heart disease, inability to establish peripheral venous access).
6. Severe cardiovascular disease, including uncontrolled hypertension, unstable angina, history of myocardial infarction within the past 6 months, congestive heart failure > NYHA (New York Heart Association) Class III, or severe arrhythmia.
7. Active infection, unexplained fever ≥ 38.5°C within 7 days prior to medication, or baseline white blood cell count > 15×10⁹/L; OR any severe acute or chronic infection requiring systemic antibacterial, antifungal, or antiviral therapy at screening (except for active hepatitis).
8. Any active autoimmune disease or history of autoimmune diseases (e.g., but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism; Patients with vitiligo; Patients with childhood asthma that has completely resolved in adulthood without any intervention are eligible; Asthma requiring bronchodilator medical intervention is excluded). Patients are eligible if: they have a history of autoimmune-related hypothyroidism and are on stable thyroid hormone replacement therapy; or have type I diabetes controlled by insulin therapy.
9. History of drug allergy.
10. Pregnant or lactating women; OR women of childbearing potential or men with pregnant partners who are unwilling to use adequate contraception during the planned trial period (from the screening visit until 120 days after the last study treatment).
11. History of organ transplantation.
12. Any other condition that, in the investigator's judgment, would make the participant unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase II Primary Outcome: Objective Response Rate (ORR) | From randomization until disease progression, assessed up to approximately 24 months
  The proportion of participants who achieve a best overall response of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
Phase I Primary Outcome: Incidence of Adverse Events (AEs) | From cell infusion up to 3 months after the last infusion
  The safety and tolerability of the autologous immune cell therapies (DC-CIK and NK) will be assessed by the incidence, type, and severity of adverse events. All AEs will be graded according to the NCI Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From the start of treatment (Phase I) or randomization (Phase II) until disease progression or death from any cause, assessed up to approximately 24 months
  The length of time during which a participant remains alive and their disease does not progress.
Overall Survival (OS) | From the start of treatment (Phase I) or randomization (Phase II) until death from any cause, assessed up to approximately 36 months
  The length of time from the start of treatment that participants are still alive.
Disease Control Rate (DCR) | From the start of treatment until the end of 4 treatment cycles, assessed up to 4 months
  The proportion of participants who achieve a best overall response of complete response (CR), partial response (PR), or stable disease (SD) according to RECIST 1.1.
Duration of Response (DoR) | From the first documented response (CR or PR) until disease progression or death, assessed up to approximately 24 months
  The length of time that a tumor continues to respond to treatment without the cancer growing or spreading.
Time to Recurrence (TTR) | From the start of treatment until disease recurrence, assessed up to approximately 24 months
  The time from the start of treatment until the first documented recurrence of the cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Minjie, Doctor, Study Chair — Liaoning Medical Diagnosis and Treatment Technology Research and Development Co., Ltd.

IPD SHARING:
Plan to Share IPD: Yes
What IPD? All of the individual participant data collected during the trial, after de-identification.
  When? Beginning 12 months after the primary publication and ending 36 months thereafter.
  With Whom? Researchers who provide a methodologically sound proposal. For What? To achieve aims in the approved proposal. Proposals should be directed to [Corresponding Author Email]. To gain access, data requestors will need to sign a data access agreement.
  Supporting Info? Study Protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF)
Supporting Information: Study Protocol
Time Frame: Beginning 12 months after the primary publication and ending 36 months thereafter.
Access Criteria: All of the individual participant data collected during the trial, after de-identification.